CLINICAL TRIAL: NCT02621476
Title: Encouraging Mail Order Pharmacy Use to Improve Outcomes and Reduce Disparities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Harvard Pilgrim Health Care (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CN-14-1947; R18DK104249 (NIH)
Record Dates: First submitted 2015-11-19; First posted 2015-12-03 (Estimated); Results first posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized intervention (Experimental): Standardized intervention to encourage mail order use and provide easily accessible information on how to access the service
  Interventions: Behavioral: Standardized intervention
- Usual care (Experimental): Usual care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Standardized intervention — Standardized intervention to encourage mail order use and provide easily accessible information on how to access the service
  Arms: Standardized intervention
Behavioral: Usual care — Usual care
  Arms: Usual care

SUMMARY:
The investigators propose a randomized encouragement trial to encourage use of the existing mail order pharmacy services among diabetes patients with poor adherence to CVD risk factor medications in 3 health care systems: Kaiser Permanente Northern California, Harvard Pilgrim, and Kaiser Permanente Hawaii.

DETAILED DESCRIPTION:
Adherence to effective cardiovascular disease (CVD) risk factor medications is associated with improved CVD risk factor control, fewer hospitalizations, and lower mortality in patients with diabetes. However, many patients are poorly adherent to medications, and there are persistent racial/ethnic and socioeconomic disparities in medication adherence. Traditional clinical trials of interventions to improve medication adherence are often resource-intensive, and focus exclusively on patient-level barriers to behavior change. Unsurprisingly, these trials have not led to sustainable, cost-effective approaches to improve adherence. Health system-level medication adherence interventions that can be implemented, "scaled up," and sustained across a wide range of health care delivery settings are urgently needed. The investigators propose a randomized encouragement trial to encourage use of existing mail order pharmacy services among diabetes patients with poor adherence to CVD risk factor medications and who only use retail pharmacies in 3 health care systems: Kaiser Permanente Northern California, Harvard Pilgrim, and Kaiser Permanente Hawaii. These combined systems include approximately 300,000 patients with diabetes with diverse racial/ethnic and socioeconomic backgrounds. Patients with no history of mail order pharmacy use will be randomized into 2 arms. In addition to examining the impact of the intervention on medication adherence and CVD risk factor control, the investigators will examine factors affecting the sustainability and dissemination of the intervention, assess the intervention's impact on utilization and health care costs, and determine whether the intervention's impact differs across racial/ethnic and socioeconomic subgroups. This research will provide a foundation for developing sustainable, system-level approaches to addressing medication adherence in diabetes patients that can be widely disseminated and implemented across a diverse array of health care systems.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes patients who are users of CVD risk factor medications (antihypertensive therapies, antihyperlipidemics therapies, and oral antihyperglycemic therapies),
* Diabetes patients considered to be poorly adherent to CVD risk factor medications within the prior 12 months
* Diabetes patients who have not used the mail order pharmacy to fill any prescribed medications at least once in the prior 12 months

Exclusion Criteria:

* Pregnancy or Dementia/Traumatic Brain Injury diagnosis in the prior 12 months
* Hospitalized, in Skilled Nursing Facility, Hospice, or Home Health at the time of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63012 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2022-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Schmittdiel, Principal Investigator — Research Scientist
Locations (1):
- Division of Research, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gregg EW, Hora I, Benoit SR. Resurgence in Diabetes-Related Complications. JAMA. 2019 May 21;321(19):1867-1868. doi: 10.1001/jama.2019.3471. No abstract available. PMID 30985875
- [Background] Lin J, Thompson TJ, Cheng YJ, Zhuo X, Zhang P, Gregg E, Rolka DB. Projection of the future diabetes burden in the United States through 2060. Popul Health Metr. 2018 Jun 15;16(1):9. doi: 10.1186/s12963-018-0166-4. PMID 29903012
- [Background] Polonsky WH, Henry RR. Poor medication adherence in type 2 diabetes: recognizing the scope of the problem and its key contributors. Patient Prefer Adherence. 2016 Jul 22;10:1299-307. doi: 10.2147/PPA.S106821. eCollection 2016. PMID 27524885
- [Background] Ho PM, Rumsfeld JS, Masoudi FA, McClure DL, Plomondon ME, Steiner JF, Magid DJ. Effect of medication nonadherence on hospitalization and mortality among patients with diabetes mellitus. Arch Intern Med. 2006 Sep 25;166(17):1836-41. doi: 10.1001/archinte.166.17.1836. PMID 17000939
- [Background] Lau DT, Nau DP. Oral antihyperglycemic medication nonadherence and subsequent hospitalization among individuals with type 2 diabetes. Diabetes Care. 2004 Sep;27(9):2149-53. doi: 10.2337/diacare.27.9.2149. PMID 15333476
- [Background] Sokol MC, McGuigan KA, Verbrugge RR, Epstein RS. Impact of medication adherence on hospitalization risk and healthcare cost. Med Care. 2005 Jun;43(6):521-30. doi: 10.1097/01.mlr.0000163641.86870.af. PMID 15908846
- [Background] Asche C, LaFleur J, Conner C. A review of diabetes treatment adherence and the association with clinical and economic outcomes. Clin Ther. 2011 Jan;33(1):74-109. doi: 10.1016/j.clinthera.2011.01.019. PMID 21397776
- [Background] Feldman R, Bacher M, Campbell N, Drover A, Chockalingam A. Adherence to pharmacologic management of hypertension. Can J Public Health. 1998 Sep-Oct;89(5):I16-8. doi: 10.1007/BF03404494. PMID 9813921
- [Background] Avorn J, Monette J, Lacour A, Bohn RL, Monane M, Mogun H, LeLorier J. Persistence of use of lipid-lowering medications: a cross-national study. JAMA. 1998 May 13;279(18):1458-62. doi: 10.1001/jama.279.18.1458. PMID 9600480
- [Background] Heisler M, Faul JD, Hayward RA, Langa KM, Blaum C, Weir D. Mechanisms for racial and ethnic disparities in glycemic control in middle-aged and older Americans in the health and retirement study. Arch Intern Med. 2007 Sep 24;167(17):1853-60. doi: 10.1001/archinte.167.17.1853. PMID 17893306
- [Background] Trinacty CM, Adams AS, Soumerai SB, Zhang F, Meigs JB, Piette JD, Ross-Degnan D. Racial differences in long-term adherence to oral antidiabetic drug therapy: a longitudinal cohort study. BMC Health Serv Res. 2009 Feb 7;9:24. doi: 10.1186/1472-6963-9-24. PMID 19200387
- [Background] Shenolikar RA, Balkrishnan R, Camacho FT, Whitmire JT, Anderson RT. Race and medication adherence in Medicaid enrollees with type-2 diabetes. J Natl Med Assoc. 2006 Jul;98(7):1071-7. PMID 16895275
- [Background] Tseng CW, Tierney EF, Gerzoff RB, Dudley RA, Waitzfelder B, Ackermann RT, Karter AJ, Piette J, Crosson JC, Ngo-Metzger Q, Chung R, Mangione CM. Race/ethnicity and economic differences in cost-related medication underuse among insured adults with diabetes: the Translating Research Into Action for Diabetes Study. Diabetes Care. 2008 Feb;31(2):261-6. doi: 10.2337/dc07-1341. Epub 2007 Nov 13. PMID 18000177
- [Background] Peeters B, Van Tongelen I, Boussery K, Mehuys E, Remon JP, Willems S. Factors associated with medication adherence to oral hypoglycaemic agents in different ethnic groups suffering from type 2 diabetes: a systematic literature review and suggestions for further research. Diabet Med. 2011 Mar;28(3):262-75. doi: 10.1111/j.1464-5491.2010.03133.x. PMID 21309834
- [Background] Duru OK, Gerzoff RB, Selby JV, Brown AF, Ackermann RT, Karter AJ, Ross S, Steers N, Herman WH, Waitzfelder B, Mangione CM. Identifying risk factors for racial disparities in diabetes outcomes: the translating research into action for diabetes study. Med Care. 2009 Jun;47(6):700-6. doi: 10.1097/mlr.0b013e318192609d. PMID 19480090
- [Background] DiMatteo MR. Variations in patients' adherence to medical recommendations: a quantitative review of 50 years of research. Med Care. 2004 Mar;42(3):200-9. doi: 10.1097/01.mlr.0000114908.90348.f9. PMID 15076819
- [Background] van Dulmen S, Sluijs E, van Dijk L, de Ridder D, Heerdink R, Bensing J. Patient adherence to medical treatment: a review of reviews. BMC Health Serv Res. 2007 Apr 17;7:55. doi: 10.1186/1472-6963-7-55. PMID 17439645
- [Background] McDonald HP, Garg AX, Haynes RB. Interventions to enhance patient adherence to medication prescriptions: scientific review. JAMA. 2002 Dec 11;288(22):2868-79. doi: 10.1001/jama.288.22.2868. PMID 12472329
- [Background] Lee JK, Grace KA, Taylor AJ. Effect of a pharmacy care program on medication adherence and persistence, blood pressure, and low-density lipoprotein cholesterol: a randomized controlled trial. JAMA. 2006 Dec 6;296(21):2563-71. doi: 10.1001/jama.296.21.joc60162. Epub 2006 Nov 13. PMID 17101639
- [Background] Duru OK, Schmittdiel JA, Dyer WT, Parker MM, Uratsu CS, Chan J, Karter AJ. Mail-order pharmacy use and adherence to diabetes-related medications. Am J Manag Care. 2010 Jan;16(1):33-40. PMID 20148603
- [Background] Schmittdiel JA, Karter AJ, Dyer W, Parker M, Uratsu C, Chan J, Duru OK. The comparative effectiveness of mail order pharmacy use vs. local pharmacy use on LDL-C control in new statin users. J Gen Intern Med. 2011 Dec;26(12):1396-402. doi: 10.1007/s11606-011-1805-7. Epub 2011 Jul 20. PMID 21773848
- [Background] Sharma KP, Taylor TN. Pharmacy effect on adherence to antidiabetic medications. Med Care. 2012 Aug;50(8):685-91. doi: 10.1097/MLR.0b013e318249d800. PMID 22354211
- [Background] Zhang L, Zakharyan A, Stockl KM, Harada AS, Curtis BS, Solow BK. Mail-order pharmacy use and medication adherence among Medicare Part D beneficiaries with diabetes. J Med Econ. 2011;14(5):562-7. doi: 10.3111/13696998.2011.598200. Epub 2011 Jul 6. PMID 21728913
- [Background] Devine S, Vlahiotis A, Sundar H. A comparison of diabetes medication adherence and healthcare costs in patients using mail order pharmacy and retail pharmacy. J Med Econ. 2010;13(2):203-11. doi: 10.3111/13696991003741801. PMID 20345227
- [Background] Fernandez EV, McDaniel JA, Carroll NV. Examination of the Link Between Medication Adherence and Use of Mail-Order Pharmacies in Chronic Disease States. J Manag Care Spec Pharm. 2016 Nov;22(11):1247-1259. doi: 10.18553/jmcp.2016.22.11.1247. PMID 27783552
- [Background] Johnsrud M, Lawson KA, Shepherd MD. Comparison of mail-order with community pharmacy in plan sponsor cost and member cost in two large pharmacy benefit plans. J Manag Care Pharm. 2007 Mar;13(2):122-34. doi: 10.18553/jmcp.2007.13.2.122. PMID 17330973
- [Background] Carroll NV, Brusilovsky I, York B, Oscar R. Comparison of costs of community and mail service pharmacy. J Am Pharm Assoc (2003). 2005 May-Jun;45(3):336-43. doi: 10.1331/1544345054003796. PMID 15991755
- [Background] Karter AJ, Parker MM, Duru OK, Schillinger D, Adler NE, Moffet HH, Adams AS, Chan J, Herman WH, Schmittdiel JA. Impact of a pharmacy benefit change on new use of mail order pharmacy among diabetes patients: the Diabetes Study of Northern California (DISTANCE). Health Serv Res. 2015 Apr;50(2):537-59. doi: 10.1111/1475-6773.12223. Epub 2014 Aug 15. PMID 25131156
- [Background] Schmittdiel JA, Marshall CJ, Wiley D, Chau CV, Trinacty CM, Wharam JF, Duru OK, Karter AJ, Brown SD. Opportunities to encourage mail order pharmacy delivery service use for diabetes prescriptions: a qualitative study. BMC Health Serv Res. 2019 Jun 25;19(1):422. doi: 10.1186/s12913-019-4250-7. PMID 31238950
- [Background] Raebel MA, Schmittdiel J, Karter AJ, Konieczny JL, Steiner JF. Standardizing terminology and definitions of medication adherence and persistence in research employing electronic databases. Med Care. 2013 Aug;51(8 Suppl 3):S11-21. doi: 10.1097/MLR.0b013e31829b1d2a. PMID 23774515
- [Background] Schmittdiel JA, Adams SR, Goler N, Sanna RS, Boccio M, Bellamy DJ, Brown SD, Neugebauer RS, Ferrara A. The impact of telephonic wellness coaching on weight loss: A "Natural Experiments for Translation in Diabetes (NEXT-D)" study. Obesity (Silver Spring). 2017 Feb;25(2):352-356. doi: 10.1002/oby.21723. PMID 28124501
- [Background] Schwab P, Racsa P, Rascati K, Mourer M, Meah Y, Worley K. A Retrospective Database Study Comparing Diabetes-Related Medication Adherence and Health Outcomes for Mail-Order Versus Community Pharmacy. J Manag Care Spec Pharm. 2019 Mar;25(3):332-340. doi: 10.18553/jmcp.2019.25.3.332. PMID 30816817
- [Background] Adams AS, Uratsu C, Dyer W, Magid D, O'Connor P, Beck A, Butler M, Ho PM, Schmittdiel JA. Health system factors and antihypertensive adherence in a racially and ethnically diverse cohort of new users. JAMA Intern Med. 2013 Jan 14;173(1):54-61. doi: 10.1001/2013.jamainternmed.955. PMID 23229831
- [Background] Liberman JN, Wang Y, Hutchins DS, Slezak J, Shrank WH. Revealed preference for community and mail service pharmacy. J Am Pharm Assoc (2003). 2011 Jan-Feb;51(1):50-7. doi: 10.1331/JAPhA.2011.09161. PMID 21247826
- [Background] Tamblyn R, Laprise R, Hanley JA, Abrahamowicz M, Scott S, Mayo N, Hurley J, Grad R, Latimer E, Perreault R, McLeod P, Huang A, Larochelle P, Mallet L. Adverse events associated with prescription drug cost-sharing among poor and elderly persons. JAMA. 2001 Jan 24-31;285(4):421-9. doi: 10.1001/jama.285.4.421. PMID 11242426
- [Background] Chernew M, Gibson TB, Yu-Isenberg K, Sokol MC, Rosen AB, Fendrick AM. Effects of increased patient cost sharing on socioeconomic disparities in health care. J Gen Intern Med. 2008 Aug;23(8):1131-6. doi: 10.1007/s11606-008-0614-0. Epub 2008 Apr 29. PMID 18443882
- [Background] Osborn CY, Cavanaugh K, Wallston KA, Kripalani S, Elasy TA, Rothman RL, White RO. Health literacy explains racial disparities in diabetes medication adherence. J Health Commun. 2011;16 Suppl 3(Suppl 3):268-78. doi: 10.1080/10810730.2011.604388. PMID 21951257
- [Background] Lewis LM, Ogedegbe C, Ogedegbe G. Enhancing adherence of antihypertensive regimens in hypertensive African-Americans: current and future prospects. Expert Rev Cardiovasc Ther. 2012 Nov;10(11):1375-80. doi: 10.1586/erc.12.138. PMID 23244358
- [Background] Schoenthaler A, Allegrante JP, Chaplin W, Ogedegbe G. The effect of patient-provider communication on medication adherence in hypertensive black patients: does race concordance matter? Ann Behav Med. 2012 Jun;43(3):372-82. doi: 10.1007/s12160-011-9342-5. PMID 22270266
- [Background] Saha S, Freeman M, Toure J, Tippens KM, Weeks C, Ibrahim S. Racial and ethnic disparities in the VA health care system: a systematic review. J Gen Intern Med. 2008 May;23(5):654-71. doi: 10.1007/s11606-008-0521-4. Epub 2008 Feb 27. PMID 18301951
- [Background] Nichols GA, Bell TJ, Pedula KL, O'Keeffe-Rosetti M. Medical care costs among patients with established cardiovascular disease. Am J Manag Care. 2010 Mar;16(3):e86-e93. PMID 20205493
- [Derived] Thomas TW, Dyer WT, Yassin M, Neugebauer R, Karter AJ, Schmittdiel JA. Is Shelter-in-Place Policy Related to Mail Order Pharmacy Use and Racial/Ethnic Disparities for Patients With Diabetes? Diabetes Care. 2021 Jun;44(6):e113-e114. doi: 10.2337/dc20-2686. Epub 2021 Apr 13. No abstract available. PMID 33849937
- [Derived] Ramachandran B, Trinacty CM, Wharam JF, Duru OK, Dyer WT, Neugebauer RS, Karter AJ, Brown SD, Marshall CJ, Wiley D, Ross-Degnan D, Schmittdiel JA. A Randomized Encouragement Trial to Increase Mail Order Pharmacy Use and Medication Adherence in Patients with Diabetes. J Gen Intern Med. 2021 Jan;36(1):154-161. doi: 10.1007/s11606-020-06237-8. Epub 2020 Oct 1. PMID 33001334
- See also: American Diabetes Association (ADA). Statistics About Diabetes — http://diabetes.org/diabetes-basics/statistics/

RESULTS

PARTICIPANT FLOW:
Groups:
- Standardized Intervention: Participants in the standardized intervention arm received outreach encouraging mail order pharmacy use.
- Control: Participants in the control arm received usual care.
Period: Overall Study
Arm/Group | Standardized Intervention | Control
Started | 31493 | 31519
Completed | 26342 | 26404
Not Completed | 5151 | 5115

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standardized Intervention | Control | Total
Number analyzed (Participants) | 31493 | 31519 | 63012
Age, Customized [Count of Participants; unit: Participants]
  <20 | 13 | 16 | 29
  20-29 | 235 | 232 | 467
  30-39 | 1323 | 1261 | 2584
  40-49 | 4429 | 4692 | 9121
  50-59 | 9198 | 9406 | 18604
  60-69 | 9132 | 9028 | 18160
  70-79 | 5092 | 4981 | 10073
  80-89 | 1890 | 1743 | 3633
  >89 | 181 | 160 | 341
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14204 | 14184 | 28388
  Male | 17289 | 17335 | 34624
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 7811 | 7815 | 15626
  Black | 3867 | 3872 | 7739
  HI/PI | 1315 | 1314 | 2629
  Asian | 5900 | 5595 | 11495
  Native American | 123 | 186 | 309
  White | 7500 | 7822 | 15322
  Missing | 4977 | 4915 | 9892
Region of Enrollment [Number; unit: participants]
  United States | 31493 | 31519 | 63012
Has Mail Order Incentive [Count of Participants; unit: Participants] | 20321 | 20007 | 40328
Has Secure Messaging [Count of Participants; unit: Participants] — This measure applies only to KPNC and KPHI participants. Population: This measure applies only to KPNC and KPHI participants.
  Participants
    number analyzed (Participants) | 26099 | 26125 | 52224
    (all) | 15009 | 15019 | 30028
Had Oral Diabetes Mellitus (DM) Drug Fill [Count of Participants; unit: Participants] | 25370 | 25400 | 50770
Had Oral Dyslipidemia (DL) Drug Fill [Count of Participants; unit: Participants] | 25924 | 25939 | 51863
Had Oral Hypertension (HT) Drug Fill [Count of Participants; unit: Participants] | 26785 | 26891 | 53676
Total Number of Oral Cardiovascular Disease (CVD) Drug Fills [Mean (Standard Deviation); unit: Oral CVD drug fills] | 13.5 (10.2) | 13.5 (10.2) | 13.5 (10.2)
Total Number of Oral HT Drug Fills [Mean (Standard Deviation); unit: Oral HT drug fills] | 7.3 (6.4) | 7.4 (6.5) | 7.4 (6.5)
Total Number of Oral DM Drug Fills [Mean (Standard Deviation); unit: Oral DM drug fills] | 5.3 (4.2) | 5.3 (4.1) | 5.3 (4.2)
# of classes of Oral CVD Drugs [Mean (Standard Deviation); unit: Classes of Oral CVD drug fills] | 3.5 (1.6) | 3.5 (1.6) | 3.5 (1.6)
# of drug classes poorly adherent to [Mean (Standard Deviation); unit: Drug classes poorly adhered to] | 1.7 (1.0) | 1.7 (1.0) | 1.7 (1.0)
% of Oral CVD drug classes poorly adherent to [Mean (Standard Deviation); unit: % of Oral CVD drug classes poorly adhere] | 57.6 (31) | 57.6 (31) | 57.6 (31)
Diabetes Identification [Count of Participants; unit: Participants]
  One Inpatient Diagnosis | 100 | 79 | 179
  One Prescription Fill | 15802 | 15760 | 31562
  Two Outpatient Diagnosis | 15591 | 15680 | 31271

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Using Mail Order Pharmacy (MOP) After Intervention
Description: users of the mail order pharmacy service - if they utilized the mail order system to deliver medications anytime in the 12 months following the date of outreach into the intervention
Time Frame: 12 months following the date of outreach into the intervention
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standardized Intervention | Control
Number analyzed (Participants) | 23642 | 26404
percentage of participants | 10.6 [10.3 to 11.0] | 9.3 [8.9 to 9.7]
Statistical Analysis 1: Comparison: Control; Test type: Superiority; p < 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: 12 months for each participant.
Arm/Group | Standardized Intervention | Control
All-Cause Mortality (participants affected / at risk) | 599/31493 | 582/31519
Serious Adverse Events (participants affected / at risk) | 0/31493 | 0/31519
Other Adverse Events (participants affected / at risk) | 0/31493 | 0/31519

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT02621476/Prot_SAP_000.pdf